CLINICAL TRIAL: NCT04313231
Title: Sterile Inflammation and Molecular Aberrations in Myelodysplastic Syndrome: Determinants of Quality of Life and Vulnerability
Brief Title: Sterile Inflammation and Molecular Aberrations in MDS
Acronym: InflamGen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: University Hospital, Bonn (Other); Universitätsklinikum Leipzig (Other)
Responsible Party: Sponsor
Other Study IDs: 20200129-2183
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: anemia; health-related quality of life; inflammation
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia; Inflammation | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDS: * Female and male patients aged 18 years and older
  * MDS, MDS/MPN diagnosis based on current WHO classification. CCUS and CHIP defined by Valent (Valent, Oncotarget, 2018) and by Stauder (Stauder, Blood, 2018)
  Interventions: Diagnostic Test: Next Generation Sequencing; Diagnostic Test: Tumorimmunological examinations - multiplex assays/quantitative polymerase chain reaction; Diagnostic Test: flow cytometry; Diagnostic Test: Metagenomics of stool samples; Diagnostic Test: Clinical/demographic data; Other: Elicitation of the HRQoL
- control: age-matched healthy persons
  Interventions: Diagnostic Test: Next Generation Sequencing; Diagnostic Test: Tumorimmunological examinations - multiplex assays/quantitative polymerase chain reaction; Diagnostic Test: flow cytometry; Diagnostic Test: Metagenomics of stool samples; Diagnostic Test: Clinical/demographic data; Other: Elicitation of the HRQoL

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing — Sequencing of patient samples will be performed in the facilities of ZIMCL. Following DNA extraction, the sequencing of granulocytes as well as of lymphocytes (control) will be carried out. IN addition to whole exome sequencing, a panel from SOPHIA GENETICS (which is also available for routine diagnostics) will be applied including the following MDS specific genes: ASXL1, BRAF, CBL, CEBPA, CSF3R, DNMT3A, EZH2, FLT3, HRAS, IDH1, IDH2, KRAS, MPL, NPM1, NRAS, RUNX1, SF3B1, SRSF2, TET2, TP53, U2AF1, WT1, ZRSR. Each patient sample will be "bulk sequenced", meaning that relevant mutations are detected down to an allele frequency of 2%.
Diagnostic Test: Tumorimmunological examinations - multiplex assays/quantitative polymerase chain reaction — Inflammasome activation is quantified by analyses of inflammasome-associated cytokine patterns. Multiplex assays for the quantification of the inflammasome-specific cytokines will be done from serum as well as from supernatants the stimulated blood cells. Cytokine quantification is carried out with Luminex FlexMap 3D. Serum cytokine levels will be quantitated in parallel.
  Quantification of RNA expression levels of inflammasome-related gene products will be performed by qPCRs from unstimulated and stimulated (=cryotube) blood cells. The necessary RNA extraction will be performed using a RNA extraction kit.
Diagnostic Test: flow cytometry — A detailed evaluation of the individual immune status is being conducted by the analysis of two specialized panels: Panel A provides a broad overview over various immune cell populations, while Panel B identifies T-cell sup-populations.
Diagnostic Test: Metagenomics of stool samples — DNA will be extracted from frozen fecal samples applying a bead-beating method using a GNOME DNA Isolation Kit (MP Biomedicals). DNA quality will be assessed using an Agilent 4200 TapeStation (Agilent Technologies). After final precipitation, DNA samples will be re-suspended in TE buffer and stored at -80 °C for further sequencing analysis. To this end, sequencing libraries will be generated using a Nextera XT DNA Sample Prep Kit (Illumina). Library quality will be confirmed using an Agilent 4200 TapeStation. Whole-genome shotgun sequencing of fecal samples will be carried out on a HiSeq2500 platform (Illumina).
Diagnostic Test: Clinical/demographic data — Demographic and clinical data include: age, age at initial diagnosis, sex, diagnosis, actual comorbidities, medication at inclusion in study, cytogenetic and molecular profiles and standard laboratory parameters (blood count, differential leukocyte count, biochemistry, iron status, inflammatory markers like CRP, albumin, fibrinogen).
Other: Elicitation of the HRQoL — Evaluation of HRQOL, of functional activities and of performance status will be done by the patient and/or the physician using validated scores.

SUMMARY:
The objective of this study is the description of the possible association between genetic mutation/aberration profiles, inflammatory tonus and clinical phenotype based on PROMs and HRQoL. Apart from gaining a better understanding of the causal correlation between genetics, sterile inflammatory processes and QoL (e.g. fatigue) in MDS, this study is supposed to identify potential novel biomarkers and, ultimately, therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients > 18 years
* MDS, MDS/MPN diagnosis based on current WHO classification. CCUS and CHIP defined by Valent (Valent, Oncotarget, 2018) and by Stauder (Stauder, Blood, 2018)
* Signed and dated declaration of consent by the patient according to ICH-GCP Guidelines

Exclusion Criteria:

* Any other illness, whether physical or mental, or any laboratory abnormalities which prevent a declaration of consent by the patient
* Patients with an acute and/or uncontrolled infection, including patients that are afebrile under treatment with antibiotic/antifungal/antiviral prophylactic medication
* Any pre-existing autoimmune disease requiring a systemic immunosuppression
* Steroid therapy (>10mg Prednison/day or equivalent), regardless of its necessity up to 4 weeks before inclusion in the study
* Anamnestic and/or current therapy with hypomethylating agents (HMA) or immunomodulatory imide drugs (IMiDs)
* Status post allogenic stem cell transplantation
* Previous or ongoing chemotherapy
* Pregnancy or breastfeeding period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MDS, MDS/MPN diagnosis based on current WHO classification. CCUS and CHIP defined by Valent (Valent, Oncotarget, 2018) and by Stauder (Stauder, Blood, 2018)
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Definition of correlation between molecular aberrations and the sterile inflammatory tonus | baseline
Definition how genetic aberrations and associated sterile inflammation impacts on health-related quality of life (HRQoL, e.g. fatigue) and functional activities in patients with MDS, MDS/MPN, or CHIP/CCUS | baseline

SECONDARY OUTCOMES:
Definition of correlation of sterile inflammatory tonus with clinical variables (e.g. progression to secondary acute myeloid leukemia (sAML), complications (e.g. infections), and survival) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Domink Wolf, Univ.Prof., Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Presentation at conferences and publication in a peer-reviewed journal

REFERENCES:
- [Background] Valent P, Stauder R, Theurl I, Geissler K, Sliwa T, Sperr WR, Bettelheim P, Sill H, Pfeilstocker M. Diagnosis, management and response criteria of iron overload in myelodysplastic syndromes (MDS): updated recommendations of the Austrian MDS platform. Expert Rev Hematol. 2018 Feb;11(2):109-116. doi: 10.1080/17474086.2018.1420473. Epub 2018 Jan 2. PMID 29292655
- [Background] Stauder R, Valent P, Theurl I. Anemia at older age: etiologies, clinical implications, and management. Blood. 2018 Feb 1;131(5):505-514. doi: 10.1182/blood-2017-07-746446. Epub 2017 Nov 15. PMID 29141943
- [Derived] Loacker L, Petzer V, Bachmann S, Griesmacher A, Wolf D, Stauder R. High concordance of clone detection between peripheral blood and bone marrow by targeted next-generation sequencing-A pilot study in patients with MDS. Br J Haematol. 2023 Aug;202(3):e16-e19. doi: 10.1111/bjh.18889. Epub 2023 Jun 1. No abstract available. PMID 37263977